CLINICAL TRIAL: NCT06151860
Title: Acute Effect of Static Stretching and Pilates Stretching on the Concentric Muscle Strength of the Knee Extensors and Flexors
Brief Title: Acute Effect of Static Stretching and Pilates Stretching on the Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do Norte do Parana (Other)
Responsible Party: Principal Investigator, Raphael Goncalves de Oliveira, Professor, Universidade Estadual do Norte do Parana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0001_UENP
Record Dates: First submitted 2023-11-17; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Muscle Strength; Muscle Strength Dynamometer
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Static stretching (Experimental): A equipment (Ladder Barrel), used in Pilates sessions, will help with the movement. To stretch the knee flexor muscles, the participant, standing, will place the dominant lower limb on the equipment and keep the other on the ground, remaining with both knees extended. The trunk will be flexed forward within the maximum range of movement achieved by the participant, until discomfort occurs in the posterior region of the thigh, but not pain. To stretch the knee extensor muscles, the participant, standing, will position the back of the foot of the dominant lower limb on the equipment and keep the other limb with the foot flat on the ground. The glute of the dominant lower limb will meet the heel of the same limb, until there is discomfort, but not pain. In both stretches, the position will be maintained for 30 seconds, followed by an equal rest time. Three series of stretching will be performed for the knee flexor muscles and then another three series for the extensor muscles.
  Interventions: Other: Static stretching
- Pilates stretching (Experimental): The protocol will be the same as the Static stretching Group, with the exception of maintaining the static position during the exercise. To do this, when stretching the knee flexor muscles, the trunk will perform continuous flexion movements until the point of muscular discomfort, followed by the extension movement, until an upright posture, continuously. On the other hand, when stretching the knee extensor muscles, the gluteal muscle of the dominant lower limb will meet the heel of the same limb, until there is discomfort, followed by the movement away, continuously.
  Interventions: Other: Pilates stretching
- Control (No Intervention)

INTERVENTIONS:
Other: Static stretching — Stretching exercises performed by maintaining the point of muscular discomfort without changing position for a certain period of time.
  Arms: Static stretching
Other: Pilates stretching — Stretching exercises performed dynamically, following the six basic principles of Pilates: concentration, control, center, precision, breathing and fluidity.
  Arms: Pilates stretching

SUMMARY:
Introduction: Studies have shown that static stretching performed immediately before strength exercises impairs performance. However, unlike static stretching, dynamic stretching performed immediately before muscular strength exercises does not seem to result in worse performance, and in some cases may even provide greater strength performance. Still, the literature is controversial and inconclusive to date.

Objective: To verify the acute effect of static stretching versus dynamic stretching on the muscle strength of young university students.

Methods: The sample will consist of 102 physically active young university students, of both sexes, aged between 18 and 25 years old, subdivided into three groups: Group 1 - static stretching; Group 2 - dynamic stretching; and Group 3 - control. Everyone will undergo assessment of the isokinetic peak torque of the knee extensor and flexor muscles at 60º/s and 180º/s in the dominant lower limb. Next, the experimental groups (Groups 1 and 2) will perform static or dynamic stretching exercises for the quadriceps and hamstring muscles, while the control group will not perform any activity. Finally, everyone will undergo muscle strength assessment again according to the same procedures used initially. Analysis of covariance (ANCOVA) will be used to compare groups, with data from the initial assessment as adjustment covariates.

ELIGIBILITY:
Inclusion Criteria:

* to practice systematic physical exercises at least three times a week over the last six months;
* healthy young adults, aged between 18 and 25 years;
* agree to participate in the study by signing the Free and Informed Consent Form.

Exclusion Criteria:

* musculoskeletal injuries in the lower limbs;
* pregnancy.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Muscle strength | Acute (immediate) effect: pre-intervention and post-intervention (10 minutes after pre-intervention)
  Concentric muscle strength of the knee extensors and flexors

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual do Norte do Paraná, Jacarezinho, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No